CLINICAL TRIAL: NCT03410017
Title: Normative Data for the Functional Listening Index - Paediatric
Brief Title: FLI Normative Study
Acronym: FLI-P
Status: Completed | Type: Observational
Sponsor: Cochlear (Industry)
Collaborators: The Hearing Cooperative Research Centre (Other); The Shepherd Centre (Unknown)
Responsible Party: Sponsor
Other Study IDs: CLTD5703
Record Dates: First submitted 2017-10-01; First posted 2018-01-25 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Hearing Loss
Keywords: Functional Listening Index
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Normally-hearing: Children with normal hearing
  Interventions: Other: Functional Listening Index

INTERVENTIONS:
Other: Functional Listening Index — Functional Listening Index questionnaire to assess acquisition of listening skills.

SUMMARY:
Single center, cross sectional observational research design to collect normative data on the acquisition of listening skills in normally-hearing children aged 0-6 years of age.

DETAILED DESCRIPTION:
The primary objective is the assessment of listening skill acquisition in normally-hearing children aged between 0 and 6 years with the Functional Listening Index - Paediatric (FLI-P). The FLI-P has been developed to address a substantial gap in the current tools available to measure the development of auditory skills in children. The FLI-P provides a measure of listening skills acquisition in children from birth to six years of age (0 - 72 months). The FLI-P will be administered by an investigator who has received appropriate training in its use or completed by parents/caregivers themselves. The FLI-P assessment will be conducted using an application running on a Personal Computer, tablet or online device. There are no specific medical or surgical procedures involved in this clinical investigation and the FLI-P is a non-interventional application.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 0 and 6 years of age.
* Pass on the Newborn Hearing Screen Status conducted during the New South Wales Statewide Infant Screening - Hearing (SWISH) Program.
* No current parental or professional concern regarding hearing status.

Exclusion Criteria:

* Pre-existing diagnosis of additional needs.
* Unrealistic expectations on the part of the subject, regarding the possible benefits, risks, and limitations of the study.
* Unwillingness or inability of the subject to comply with all investigational requirements.

Ages: 1 Day to 6 Years | Sex: All
Age Groups: Child
Study Population: Up to 700 normally-hearing children aged between 0 to 6 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 536 (Actual)
Dates: Start 2017-11-03 (Actual); Primary Completion 2018-10-08 (Actual); Study Completion 2018-12-17 (Actual)

PRIMARY OUTCOMES:
Functional Listening Index | 1 day
  The assessment of listening skill acquisition in normally-hearing children aged between 0 and 6 years with the Functional Listening Index - Paediatric (FLI-P).

CONTACTS AND LOCATIONS:
Overall Officials: Aleisha Davis, MLSP, Principal Investigator — The Hearing Cooperative Research Centre
Locations (1):
- The MARCS Institute Western Sydney University, Milperra, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-07): https://cdn.clinicaltrials.gov/large-docs/17/NCT03410017/Prot_SAP_000.pdf